CLINICAL TRIAL: NCT00949520
Title: Dual Source Computed Tomography (DSCT) During Injection of Dipyridamole : a New Technique for Myocardial Ischemia Assessment
Brief Title: Stress Multidetector Computed Tomography (MDCT) an New Diagnostic Tool for Myocardial Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009/12; 2009-A00364-53
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Coronary Artery Lesion
Keywords: patients; functional evaluation; known coronary artery lesion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: coronary dual source computed tomography (DSCT) — coronary dual source computed tomography during dipyridamole injection
  Other Names: coronary DSCT
Other: myocardial single photon emission computed topography (SPECT) — myocardial single photon emission computed topography during dipyridamole injection
  Other Names: myocardial SPECT

SUMMARY:
The goal of this study is to evaluate the ability of MDCT under stress to assess myocardial ischemia. There is some preliminary data in the literature showing the ability of MDCT under stress to bring relevant information about myocardial ischemia. Stress MDCT will have several advantages over single photon emission computed tomography (SPECT) imaging namely: shorter acquisition time, lower irradiation dose, lower cost. The feasibility of such experiment is still debated and need to be address in a clinical study.

DETAILED DESCRIPTION:
Hypothesis: Cardiac dual source computed tomography (DSCT) performed during dipyridamole infusion allows for 1) myocardial perfusion analysis and detection of myocardial ischemia and 2) good quality evaluation (artefact free) of the coronary artery anatomy. Cardiac DSCT during dipyridamole infusion may assess in a single volume acquisition relevant information about coronary anatomy and myocardial ischemia that required today two different examinations each with a cost and side effects. Recently investigators showed on animal models as well as in humans that MDCT during stress test could detect myocardial ischemia.

Purposes: 1) To evaluate the diagnostic potential sensitivity, specificity of coronary DSCT during dipyridamole infusion for the assessment of myocardial ischemia with myocardial single photon emission computed topography (SPECT) as standard of reference. 2) To evaluate the feasibility (presence of artefact, number of coronary segment assessable) of coronary DSCT during dipyridamole injection.

Methods: This prospective study will include patients referred from the department of cardiology of Nord hospital. Inclusion criteria will be: patients who required functional evaluation of a known coronary artery lesion. Patients will be successively include. Each patient will undergo myocardial SPECT and coronary DSCT during dipyridamole injection. Coronary DSCT image analysis will determine the severity and the extension of the ischemic territory. Statistical analysis will determine the reproductibility of the described technique, compared the DSCT with SPECT as standard of reference and determined sensitivity, specificity and predictive values (positive and negative) of the described technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients who required functional evaluation of a known coronary artery lesion

Exclusion Criteria:

* Disorders of the heart rhythm
* Myocardial infarct dating less than a month
* Unstable anger
* Congestive heart failure stages 3 and 4 of NYHA
* Renal failure
* Pregnancy and feeding
* History of anaphylactic reaction in the injection of iodized product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-07; Primary Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the diagnostic potential sensitivity, specificity of coronary DSCT during dipyridamole infusion for the assessment of myocardial ischemia with myocardial single photon emission computed topography (SPECT) as standard of reference. | 1 year

SECONDARY OUTCOMES:
To evaluate the feasibility (presence of artefact, number of coronary segment assessable) of coronary DSCT during dipyridamole injection. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Jacquier, Principal Investigator — Assistance Publique-Hôpitaux de Marseille
Locations (1):
- Assistance Publique-Hôpitaux de Marseille, Marseille, France